CLINICAL TRIAL: NCT01573858
Title: Effect of Acupuncture and Clomiphene Citrate on Live Birth in Anovulatory Women With Polycystic Ovary Syndrome: A Randomized Controlled Trial (PCOSAct)
Brief Title: Acupuncture and Clomiphene Citrate on Live Birth in Anovulatory Women With Polycystic Ovary Syndrome
Acronym: PCOSAct
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Collaborators: Yale University (Other); Penn State University (Other); Göteborg University (Other); The University of Hong Kong (Other); Beijing University of Chinese Medicine (Other); Sichuan University (Other); Second Affiliated Hospital of Heilongjiang University of Chinese Medicine (Other); Harbin Medical University (Other); Daqing Oil Field Hospital (Other); Daqing Longnan Hospital (Unknown); Liaoning University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine (Other); Tianjin Tanggu Maternity and Child Care Center (Unknown); Wenzhou Chinese Medicine Hospital (Unknown); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Hangzhou Chinese Medicine Hospital (Unknown); Shanxi Chinese Medicine Hospital (Unknown); Henan Chinese Medicine Hospital (Unknown); Maternal and Child Health Hospital of Xuzhou (Unknown); Huaian Maternal and Child Health Care Hospital (Other); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other); Suzhou Chinese Medicine Hospital (Unknown); Wuhan TongJi Hospital (Other); Hubei Chinese Medicine Hospital (Unknown); Jiangxi University of Chinese Medicine Affiliated Hospital (Unknown); The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Guangdong Provincial People's Hospital (Other); Guangzhou Liwan Chinese Hospital (Unknown); Dalian maternity hospital (Unknown)
Responsible Party: Principal Investigator, Xiaoke Wu, Professor and Department Chairman of Obstetrics and Gynecology, Heilongjiang University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCOSAct
Record Dates: First submitted 2012-04-04; First posted 2012-04-10 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Pregnancy; Polycystic Ovary Syndrome; Infertility
Keywords: Infertility; Polycystic Ovary Syndrome; Clomiphene citrate; Acupuncture
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Acupuncture treatment 1 plus CC (Experimental)
  Interventions: Other: Acupuncture treatment 1; Other: CC
- Acupuncture treatment 2 plus CC (Active Comparator)
  Interventions: Other: Acupuncture treatment 2; Other: CC
- Acupuncture treatment 1 plus CC placebo (Active Comparator)
  Interventions: Other: Acupuncture treatment 1; Other: CC placebo
- Acupucture treatment 2 and CC placebo. (Active Comparator)
  Interventions: Other: Acupuncture treatment 2; Other: CC placebo

INTERVENTIONS:
Other: Acupuncture treatment 1 — Two sets of acupuncture points will be alternated every second treatment. The first set consists of CV3, CV 6, and ST 29 bilaterally，SP 6 and SP 9 bilaterally. Needles will also be placed in LI bilaterally and GV 20. CV 3, CV 6, ST 29, SP 6, and SP 9 will be connected to and electrical stimulator and stimulated with low-frequency EA of 2Hz, 0.3 ms.
  Arms: Acupuncture treatment 1 plus CC; Acupuncture treatment 1 plus CC placebo
Other: Acupuncture treatment 2 — Needles will be inserted to a depth of <5 mm, one in each shoulder and on in each upper arm at non-acupuncture points. Electrodes will be attached to the needles and the stimulator will be turned on at an intensity of zero (no active current) in order to mimic EA in the acupuncture treatment 1. No manual stimulation of the needles will be performed.
  Arms: Acupucture treatment 2 and CC placebo.; Acupuncture treatment 2 plus CC
Other: CC — CC 50 mg every day for 5 days (day 3-7 of cycle), for a total of 4 cycles. Non-response will be defined after 4 weeks of CC placebo administration with 3 consecutive weekly negative P4 and hCG levels. Then during the fifth week a higher dose consisting of one more tablet per day (up to 3 tablets per day at third or fourth cycles, if they remain non-responders) will be given 5 days.
  Arms: Acupuncture treatment 1 plus CC; Acupuncture treatment 2 plus CC
Other: CC placebo — CC placebo 50 mg every day for 5 days (day 3-7 of cycle), for a total of 4 cycles. Non-response will be defined after 4 weeks of CC Placebo administration with 3 consecutive weekly negative P4 and hCG levels. Then during the fifth week a higher dose consisting of one more tablet per day (up to 3 tablets per day at third or fourth cycles, if they remain non-responders) will be given 5 days.
  Arms: Acupucture treatment 2 and CC placebo.; Acupuncture treatment 1 plus CC placebo

SUMMARY:
The objectives of the present trial are to test the following three hypotheses in anovulatory women with PCOS:

1. Acupuncture protocol 1 plus CC (Arm A) is more likely to result in live birth than acupuncture protocol 2 combined with CC (Arm B),
2. Acupuncture protocol 2 plus CC (Arm B) is more likely to result in live birth than acupuncture protocol 1 plus placebo (Arm C),
3. Acupuncture protocol 1 plus placebo (Arm C) is more likely to result in live birth than acupuncture protocol 2 plus placebo (Arm D).

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled, 2 by 2 factorial clinical trial for Chinese women with PCOS.

Primary outcomes:

- Live birth rate

Secondary outcomes:

* Ovulation rate
* Ongoing pregnancy rate
* Multiple pregnancy rate
* Miscarriage rate
* Hormonal profile
* Metabolic profile
* Side effect profile

ELIGIBILITY:
1. Inclusion Criteria:

   * Age of women between 20 and 40 years.
   * Confirmed diagnosis of PCOS according to the modified Rotterdam criteria and all subjects must have anovulation plus either polycystic ovaries and/or hyperandro-genism.
   * Patency of at least one tube and a normal uterine cavity shown by hysterosalpingogram, HyCosi or diagnostic laparoscopy.
   * Semen analysis:

     1. a. Sperm concentration ≥15×106/ml and b. total motility (a+b+c) ≥40% or forward motility (a+b) ≥32% in the semen analysis of the husband (based on World Health Organization, 2010).
     2. Total motile sperm count ≥9 million [based on WHO (2010) criteria, volume 1.5 ml; conc 15 million; motility 40%. 1.5 x 15 x 0.04=9 million].
2. Exclusion Criteria:

   * Exclusion of other endocrine disorders

     * Patients with hyperprolactinemia (defined as two prolactin levels at least one week apart 25 ng/mL or greater or as determined by local normative values). The goal of eliminating patients with documented hyperprolactinemia is to decrease the heterogeneity of the PCOS population. These patients may be candidates for ovulation induction with alternate regimens (dopamine agonists). A normal level within the last year or on treatment is adequate for entry.
     * Patients with FSH levels > 15 mIU/mL. A normal level within the last year is adequate for entry.
   * Patients with uncorrected thyroid disease (defined as TSH < 0.2 mIU/mL or > 5.5 mIU/mL). A normal level within the last year is adequate for entry.

     * Patients diagnosed with Type I or Type II diabetes who are poorly controlled (defined as a glycohemoglobin level > 7.0%), or patients receiving antidiabetic medications such as insulin, thiazolidinediones, acarbose, or sulfonylureas likely to confound the effects of study medication; patients currently receiving metformin XR for a diagnosis of Type I or Type II diabetes or for PCOS are also specifically excluded.
     * Patients with suspected Cushing's syndrome.
   * Use of hormonal or other medication including Chinese Herbal prescriptions which may affect the outcome at least in the past 2 months.
   * Pregnancy within the past 6 weeks.
   * Within 6 weeks post-abortion or postpartum.
   * Breastfeeding within the last 6 months.
   * Acupuncture within the last 6 months.
   * Not willing to give written consent to the study.
   * Additional exclusion criteria

     * Patients on oral contraceptives, depot progestins, or hormonal implants (including Implanon). A two month washout period will be required prior to screening for patients on these agents. Longer washouts may be necessary for certain depot contraceptive forms or implants, especially where the implants are still in place. A one-month washout will be required for patients on oral cyclic progestins.
     * Patients with liver disease defined as AST or ALT > 2 times normal or total bilirubin >2.5 mg/dL. Patients with renal disease defined as BUN > 30 mg/dL or serum creatinine> 1.4 mg/dL.
     * Patients with significant anemia (Hemoglobin < 10 g/dL).
     * Patients with a history of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident.
     * Patients with known heart disease that is likely to be exacerbated by pregnancy.
     * Patients with a history of, or suspected cervical carcinoma, endometrial carcinoma, or breast carcinoma. A normal Pap smear result will be required for women 21 and over.
     * Patients with a current history of alcohol abuse. Alcohol abuse is defined as > 14 drinks/week or binge drinking.
     * Patients enrolled simultaneously into other investigative studies that require medications, proscribe the study medications, limit intercourse, or otherwise prevent compliance with the protocol.
     * Patients who anticipate taking longer than a one month break during the protocol should not be enrolled.
     * Patients taking other medications known to affect reproductive function or metabolism. These medications include oral contraceptives, GnRH agonists and antagonists, antiandrogens, gonadotropins, anti-obesity drugs, Chinese herbal formula, anti-diabetic drugs such as metformin and thiazolidinediones, somatostatin, diazoxide, ACE inhibitors, and calcium channel blockers. The washout period on all these medications will be two months.
     * Patients with a suspected adrenal or ovarian tumor secreting androgens.
     * Couples with previous sterilization procedures (vasectomy, tubal ligation) which have been reversed. The prior procedure may affect study outcomes, and patients with both a reversed sterilization procedure and PCOS are rare enough that exclusion should not adversely affect recruitment.
     * Subjects who have undergone a bariatric surgery procedure in the recent past (< 12 months) and are in a period of acute weight loss or have been advised against pregnancy by their bariatric surgeon.
     * Patients with untreated poorly controlled hypertension defined as a systolic blood pressure 160 mm Hg or a diastolic 100 mm Hg obtained on two measures obtained at least 60 minutes apart.
     * Patients with known congenital adrenal hyperplasia.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2012-07-06 (Actual); Primary Completion 2014-11-08 (Actual); Study Completion 2015-10-07 (Actual)

PRIMARY OUTCOMES:
Live birth rate | Up to 3 years

SECONDARY OUTCOMES:
Ovulation rate | Up to 3 years
Ongoing pregnancy rate | Aprial 2012 to July 2014 (up to 3 years)
  Up to 3 years
Multiple pregnancy rate | Up to 2 years
Miscarriage rate | Up to 2 years
  loss of an intrauterine pregnancy before 20 completed weeks of gestation.
Hormonal profile | Up to 2 years
  Hormonal profile include: Testosterone(T), Sex hormone-binding globulin (SHBG), Follicle stimulating hormone (FSH),Luteinizing hormone(LH),and Dehydroepiandrosterone sulfate (DHEAS).
Metabolic profile | Up to 2 years
  Metabolic profile includes: Serum glucose concentration, Insulin concentration, cholesterol, Triglycerides (TG), High density lipoprotein cholesterol (HDL-C) and Low density lipoprotein cholesterol (LDL-C)
Side effect profile | Up to 2 years
  Side effects of CC include hot flashes, mood changes, bloating, formation of ovarian cysts, and pain, extremely rare are pituitary apoplexy and deep venous thrombosis. The major side effects of acupuncture are local skin irritation, discomfort, and vasovagal reactions during the procedure. All above mentioned side effects will be recorded weekly.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoke Wu, M.D., Ph.D., Principal Investigator — First Affiliated Hospital of Heilongjiang Chinese Medicine University; Lihui Hou, M.D., Principal Investigator — First Affiliated Hospital of Heilongjiang Chinese Medicine University; Richard Legro, MD, Study Chair — Steering Committee, Pennsylvania State University College of Medicine; Heping Zhang, PHD, Study Chair — Data and Quality Control, Yale University
Locations (25):
- China (25):
  - First Affiliated Hospital，Anhui University of Chinese Medicine, Hefei, Anhui
  - First Affiliated Hospital，Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Guangzhou Liwan Chinese Hospital, Guangzhou, Guangdong
  - Guangdong Chinese Hospital, Guangzhou, Guangdong
  - Daqing LongNa Hospital, Daqing, Heilongjiang
  - The Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Forth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Second Affiliated Hospital，Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - First Affiliated Hospital，Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - Henan Chinese Medicine Hospital, Zhengzhou, Henan
  - Wuhan Tongji Hospital, Wuhan, Hubei
  - Hubei Chinese Medicine Hospital, Wuhan, Hubei
  - First Affiliated Hospital，Hunan University of Chinese Medicine, Changsha, Hunan
  - Maternal and Child Health Hospital of Huaian, Huaian, Jiangsu
  - Suzhou Chinese Medicine Hospital, Suzhou, Jiangsu
  - Maternal and Child Health Hospital of Xuzhou, Xuzhou, Jiangsu
  - Jiangxi University of Chinese Medicine Affiliated Hospital, Nanchang, Jiangxi
  - Dalian maternity hospital, Dalian, Liaoning
  - Liaoning University of Chinese Medicine Affiliated Hospital, Shenyang, Liaoning
  - Shanxi Chinese Medicine Hospital, Shangxi, Shanxi
  - First Affiliated Hospital，Tianjin University of Chinese Medicine, Tianjin, Tianjin Municipality
  - Tianjin Tanggu Maternity and Child Care Center, Tianjin, Tianjin Municipality
  - Integrated Chinese and Western Medicine Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Wenzhou Chinese Medicine Hospital, Wenzhou, Zhejiang
  - Hangzhou Chinese Medicine Hospital, Hangzhou

REFERENCES:
- [Derived] Li J, Wu Q, Cong J, Chang H, Ma HL, Zhang DJ, Wang Y, Zhang RZ, Kam RKT, Ho CS, Chan MHM, Ma RCW, Ng EHY, Mol BWJ, Stener-Victorin E, Legro RS, Wang CC, Wu XK; PCOSAct Study Group. Total Testosterone Measured by Liquid Chromatograph-Tandem Mass Spectrometry Refines Diagnosis of Biochemical Hyperandrogenism and Better Identifies Subgroup at Genuine Risk of Adverse Fertility Outcomes in Women With Polycystic Ovary Syndrome. Reprod Med Biol. 2026 Jan 28;25(1):e70013. doi: 10.1002/rmb2.70013. eCollection 2026 Jan-Dec. PMID 41613610
- [Derived] Gong Y, Li J, Ma HL, Jiang T, Qin HC, Li MB, Wu XK. High acupuncture expectancy is associated with shorter time to ovulation and higher chances of ovulation in infertile patients with PCOS receiving acupuncture: a secondary analysis of a randomized controlled trial. Acupunct Med. 2025 Jun;43(3):137-143. doi: 10.1177/09645284251342261. Epub 2025 May 19. PMID 40390321
- [Derived] Chang H, Shi B, Ge H, Liu C, Wang L, Ma C, Liu L, Zhang W, Zhang D, Wang Y, Wang CC, Wu X. Acupuncture improves the emotion domain and lipid profiles in women with polycystic ovarian syndrome: a secondary analysis of a randomized clinical trial. Front Endocrinol (Lausanne). 2023 Aug 29;14:1237260. doi: 10.3389/fendo.2023.1237260. eCollection 2023. PMID 37711905
- [Derived] Luo X, Yang XM, Cai WY, Chang H, Ma HL, Peng Y, Wu XK. Decreased Sex Hormone-Binding Globulin Indicated Worse Biometric, Lipid, Liver, and Renal Function Parameters in Women with Polycystic Ovary Syndrome. Int J Endocrinol. 2020 Jun 25;2020:7580218. doi: 10.1155/2020/7580218. eCollection 2020. PMID 33101409
- [Derived] Zhang D, Gao J, Liu X, Qin H, Wu X. Effect of Three Androgen Indexes (FAI, FT, and TT) on Clinical, Biochemical, and Fertility Outcomes in Women with Polycystic Ovary Syndrome. Reprod Sci. 2021 Mar;28(3):775-784. doi: 10.1007/s43032-020-00316-1. Epub 2020 Sep 28. PMID 32989632
- [Derived] Zhang D, Yang X, Li J, Yu J, Wu X. Effect of hyperinsulinaemia and insulin resistance on endocrine, metabolic and fertility outcomes in women with polycystic ovary syndrome undergoing ovulation induction. Clin Endocrinol (Oxf). 2019 Sep;91(3):440-448. doi: 10.1111/cen.14050. Epub 2019 Jun 28. PMID 31222771
- [Derived] Ma HL, Xie LZ, Gao JS, Cong J, Deng YY, Ng EHY, Liu JP, Wu XK. Acupuncture and clomiphene for Chinese women with polycystic ovary syndrome (PCOSAct): statistical analysis approach with the revision and explanation. Trials. 2018 Nov 1;19(1):601. doi: 10.1186/s13063-018-2942-7. PMID 30382872
- [Derived] Li J, Wu Q, Wu XK, Zhou ZM, Fu P, Chen XH, Yan Y, Wang X, Yang ZW, Li WL, Stener-Victorin E, Legro RS, Ng EH, Zhang H, Mol BWJ, Wang CC; for PCOSAct Study Group. Effect of exposure to second-hand smoke from husbands on biochemical hyperandrogenism, metabolic syndrome and conception rates in women with polycystic ovary syndrome undergoing ovulation induction. Hum Reprod. 2018 Apr 1;33(4):617-625. doi: 10.1093/humrep/dey027. PMID 29471520
- [Derived] Wu XK, Stener-Victorin E, Kuang HY, Ma HL, Gao JS, Xie LZ, Hou LH, Hu ZX, Shao XG, Ge J, Zhang JF, Xue HY, Xu XF, Liang RN, Ma HX, Yang HW, Li WL, Huang DM, Sun Y, Hao CF, Du SM, Yang ZW, Wang X, Yan Y, Chen XH, Fu P, Ding CF, Gao YQ, Zhou ZM, Wang CC, Wu TX, Liu JP, Ng EHY, Legro RS, Zhang H; PCOSAct Study Group. Effect of Acupuncture and Clomiphene in Chinese Women With Polycystic Ovary Syndrome: A Randomized Clinical Trial. JAMA. 2017 Jun 27;317(24):2502-2514. doi: 10.1001/jama.2017.7217. PMID 28655015